CLINICAL TRIAL: NCT02917096
Title: Pilot Open-Label Study of Safety and Efficacy of Ruxolitinib Given Peri-Transplant During Reduced Intensity Allogeneic Hematopoietic Cell Transplantation (HCT) in Patients With Myelofibrosis
Brief Title: Ruxolitinib Phosphate and Chemotherapy Given Before and After Reduced Intensity Donor Stem Cell Transplant in Treating Patients With Myelofibrosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16337; NCI-2016-01400 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 16337 (Other: City of Hope Medical Center)
Record Dates: First submitted 2016-09-26; First posted 2016-09-28 (Estimated); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Primary Myelofibrosis; Secondary Myelofibrosis
MeSH Terms: conditions — Primary Myelofibrosis | interventions — fludarabine; fludarabine phosphate; Melphalan; ruxolitinib; Sirolimus; Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (ruxolitinib phosphate, chemotherapy,allogeneic HCT) (Experimental): PREPARATIVE REGIMEN: Patients receive fludarabine phosphate IV on days -9 to -5, melphalan IV over 20 minutes on day -4, and ruxolitinib phosphate PO BID on days -3 to 30 with a taper for 2-3 weeks in the absence of disease progression or unacceptable toxicity. Patients being treated with ruxolitinib phosphate prior to allogeneic HCT as standard therapy may continue receiving ruxolitinib phosphate.
  GVHD PROPHYLAXIS: Patients receive tacrolimus IV continuously beginning on day -3 and convert to PO daily when the patient is able to tolerate and absorb oral medications. Patients also receive sirolimus PO daily beginning on day -3. Treatment continues in the absence of GVHD.
  STEM CELL TRANSPLANT: Patients undergo allogeneic HCT on day 0.
  Interventions: Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Drug: Fludarabine; Drug: Fludarabine Phosphate; Other: Laboratory Biomarker Analysis; Drug: Melphalan; Other: Pharmacological Study; Drug: Ruxolitinib; Drug: Ruxolitinib Phosphate; Drug: Sirolimus; Drug: Tacrolimus

INTERVENTIONS:
Procedure: Allogeneic Hematopoietic Stem Cell Transplantation — Undergo allogeneic HCT
  Other Names: Allogeneic Hematopoietic Cell Transplantation; Allogeneic Stem Cell Transplantation; HSC; HSCT
Drug: Fludarabine — Given IV
  Other Names: Fluradosa
Drug: Fludarabine Phosphate — Given IV
  Other Names: 2-F-ara-AMP; 9H-Purin-6-amine, 2-fluoro-9-(5-O-phosphono-.beta.-D-arabinofuranosyl)-; Beneflur; Fludara; SH T 586
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Melphalan — Given IV
  Other Names: Alanine Nitrogen Mustard; CB-3025; L-PAM; L-Phenylalanine Mustard; L-sarcolysin; L-Sarcolysin Phenylalanine mustard; L-Sarcolysine; Melphalanum; Phenylalanine Mustard; Phenylalanine nitrogen mustard; Sarcoclorin; Sarkolysin; WR-19813
Other: Pharmacological Study — Correlative studies
Drug: Ruxolitinib — Given PO
  Other Names: INCB-18424; INCB18424; Oral JAK Inhibitor INCB18424
Drug: Ruxolitinib Phosphate — Given PO
  Other Names: INCB-18424 Phosphate; Jakafi
Drug: Sirolimus — Given PO
  Other Names: AY 22989; RAPA; Rapamune; Rapamycin; SILA 9268A; WY-090217
Drug: Tacrolimus — Given IV and PO
  Other Names: FK 506; Fujimycin; Hecoria; Prograf; Protopic

SUMMARY:
This pilot clinical trial studies the side effects and best dose of ruxolitinib phosphate when given together with chemotherapy before and after a donor stem cell transplant in treating patients with myelofibrosis. Ruxolitinib phosphate may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as fludarabine phosphate and melphalan, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving ruxolitinib phosphate together with chemotherapy before and after a donor stem cell transplant may help stop the growth of cells in the bone marrow, including normal blood-forming cells (stem cells) and cancer cells. It may also stop the patient's immune system from rejecting the donor's stem cells. When the healthy stem cells from a donor are infused into the patient they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets. The donated stem cells may also replace the patient?s immune cells and help destroy any remaining cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Among the dose levels tested, to determine the maximum tolerated dose (MTD) and recommended phase II dose (RP2D) of ruxolitinib phosphate (ruxolitinib), when given as part of reduced intensity allogeneic hematopoietic cell transplant (HCT), in patients with myelofibrosis.

II. To determine if the addition of ruxolitinib is safe by evaluation of toxicities including: type, frequency, severity, attribution, time course and duration.

SECONDARY OBJECTIVES:

I. To characterize and evaluate hematologic recovery, donor cell engraftment and immune reconstitution by cell count and flow cytometry of lymphocyte subsets.

II. To estimate the cumulative incidence of acute graft-versus-host disease (aGVHD) and non-relapse mortality (NRM) at 100-days post transplant.

III. To estimate the cumulative incidence of chronic GVHD at 1- and 2-years post transplant.

IV. To estimate the probabilities of overall and progression-free survival (OS/PFS) at 1- and 2-years post transplant.

V. To characterize changes in aGVHD biomarkers (Reg-3 alpha, soluble tumor necrosis factor receptor I [sTNF RI], IL2R alpha), janus associated kinases (JAK)-regulated pro-inflammatory cytokines (i.e. IL-6, TNF alpha, CRP, beta 2microglobulin) and STAT3 phosphorylation (downstream of JAK signaling) over time and by aGVHD status/grade.

OUTLINE: This is a dose-escalation study of ruxolitinib phosphate.

PREPARATIVE REGIMEN: Patients receive fludarabine phosphate intravenously (IV) on days -9 to -5, melphalan IV over 20 minutes on day -4, and ruxolitinib phosphate orally (PO) twice daily (BID) on days -3 to 30 with a taper for 2-3 weeks in the absence of disease progression or unacceptable toxicity.

GVHD PROPHYLAXIS: Patients receive tacrolimus IV continuously beginning on day -3 and convert to PO daily when the patient is able to tolerate and absorb oral medications. Patients also receive sirolimus PO daily beginning on day -3. Treatment continues in the absence of GVHD.

STEM CELL TRANSPLANT: Patients undergo allogeneic HCT on day 0.

After completion of study treatment, patients are followed up for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Primary or secondary myelofibrosis intermediate or high risk by Dynamic International Prognostic Scoring System (DIPSS) in chronic or accelerated phase
* Performance status of >= 70% on the Karnofsky scale
* The effects of chemotherapy, ruxolitinib on the developing fetus are unknown; for this reasonWomen of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control or abstinence) prior to study entry and for 1 year following transplant as per City of Hope standard operating procedure (SOP) for allogeneic transplantation; should a woman become pregnant or suspect that she is pregnant while participating on the trial, she should inform her treating physician immediately
* Bone marrow and peripheral blood studies must be available for confirmation of diagnosis; cytogenetics, flow cytometry, and molecular studies (such as JAK-2, MPL and CALR mutational status) will be obtained as per standard practice
* Bone marrow aspirates/biopsies should be performed within 30 +/- 3 days from registration to confirm disease remission status
* All candidates for this study must have a human leukocyte antigen (HLA) (A, B, C, DR) identical siblings who is willing to donate bone marrow for primed blood stem cells or an 8/8 allele-matched unrelated donor
* All ABO blood group combinations of the donor/recipient are acceptable since even major ABO compatibilities can be dealt with by various techniques (red cell exchange or plasma exchange)
* A cardiac evaluation with an electrocardiogram showing no ischemic changes or abnormal rhythm and an ejection fraction of 50% established by multi-gated acquisition scan (MUGA) or echocardiogram
* Patients must have creatinine of less than or equal to 1.5 mg/dL or creatinine clearance > 60 ml/min
* A bilirubin of up to 2.0 mg/dL, excluding patients with Gilbert's disease
* Patients should also have a serum glutamic oxaloacetic transaminase (SGOT) and serum glutamate pyruvate transaminase (SGPT) less than 5 times the upper limit of normal
* Pulmonary function test including diffusion capacity of the lung for carbon monoxide (DLCO) will be performed; forced expiratory volume in 1 second (FEV1) and DLCO should be greater than 50% of predicted normal value
* All subjects must have the ability to understand and the willingness to sign a written informed consent that has been approved by the City of Hope Institutional Review Board (COH IRB); the patient, a family member and transplant staff physician (physician, nurse, social worker) will meet at least once prior to the subject signing consent; during this meeting all pertinent information with respect to risks and benefits to donor and recipient will be presented; alternative treatment modalities will be discussed; the risks are explained in detail in the enclosed consent form
* Prior therapy with hydroxyurea, interferon, anagrelide, ruxolitinib, hypomethylating agents, revlimid, thalidomide, steroids, other JAK inhibitors is allowed; for acute myeloid leukemia (AML) patients who are back in chronic phase myeloproliferative neoplasm (MPN), prior induction therapy is allowed

Exclusion Criteria:

* Patients should not have any uncontrolled illnesses including ongoing or active infection
* Patients may not be receiving any other investigational agents, or concurrent biological, chemotherapy, or radiation therapy
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to ruxolitinib
* Pregnant women are excluded from this study because ruxolitinib is an agent with the potential for teratogenic or abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with ruxolitinib, breastfeeding should be discontinued if the mother is treated with ruxolitinib
* Patients with active 2nd malignancies other than myelofibrosis, AML, excised skin cancer, early stage cervical and prostate cancer
* Previous allogeneic hematopoietic stem cell transplantation
* Any psychiatric, social or compliance issues that, in the treating physician opinion, will interfere with completion of the transplant treatment and follow up
* Patients who have been treated with chemotherapy or radiation within two weeks of planned study enrollment; this does not include hydroxyurea, which may be continued until start of conditioning therapy; ruxolitinib may be continued at principal investigator's discretion during conditioning
* Non-compliance; defined as any subject, who in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2016-11-13 (Actual); Primary Completion 2020-04-16 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of ruxolitinib phosphate, defined as less than or equal to 1 of 6 dose limiting toxicities, graded according to the Bearman criteria and the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.03 | Up to 45 days post stem cell infusion
  Will be summarized in terms of type (organ affected, or laboratory determination) severity, time of onset, duration, probable associates with the study treatment and reversibility or outcome.

SECONDARY OUTCOMES:
Engraftment (recovery of granulopoiesis and megakaryopoiesis) | Up to 100 days post stem cell infusion
  Defined as absolute neutrophil count >= 0.5 x 10^3/ul sustained for 3 consecutive lab values on different days with no subsequent decline, and platelets >= 20 K/ul independent of platelet transfusion support.
Cumulative incidence of acute graft-versus-host disease (aGVHD), graded and staged according to the Consensus Grading | Up to 100 days post stem cell infusion
  Will be calculated using the Gray method with prior death or relapse considered competing events.
Cumulative incidence of chronic GVHD, graded and staged according to the Consensus Grading | Up to 100 days post stem cell infusion
  Will be calculated using the Gray method with prior death or relapse considered competing events.
Incidence of infections | Up to 100 days post stem cell infusion
  Will be reported by site of disease, date of onset, severity and resolution, if any.
Overall survival | From the day of stem cell infusion until death, or last follow-up, whichever occurs first, assessed for up to 2 years
  Will be calculated using the Kaplan-Meier method.
Progression-free survival | From the day of stem cell infusion to the date of death, disease relapse/progression, or last follow-up, whichever occurs first, assessed for up to 2 years
  Will be calculated using the Kaplan-Meier method.
Cumulative incidence of relapse/progression | Up to 2 years
  Will be calculated as a competing risk using the Gray method.
Non-relapse mortality, defined as death occurring in a patient from causes other than relapse or progression | Up to 2 years
  Will be calculated as a competing risk using the Gray method.

CONTACTS AND LOCATIONS:
Overall Officials: Haris Ali, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States

REFERENCES:
- [Derived] Ali H, Tsai NC, Synold T, Mokhtari S, Tsia W, Palmer J, Stiller T, Al Malki M, Aldoss I, Salhotra A, Rahmanuddin S, Pullarkat V, Cai JL, Stein A, Forman SJ, Marcucci G, Mei M, Snyder DS, Nakamura R. Peritransplantation ruxolitinib administration is safe and effective in patients with myelofibrosis: a pilot open-label study. Blood Adv. 2022 Mar 8;6(5):1444-1453. doi: 10.1182/bloodadvances.2021005035. PMID 34581764